CLINICAL TRIAL: NCT05413889
Title: Validation and Implementation Design of a Pragmatic Randomized Controlled Trial Leveraging Epic Systems 30-day Unplanned Readmission Risk Model
Brief Title: Validation and Implementation Design of an Epic Systems 30-day Unplanned Readmission Risk Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00079395
Record Dates: First submitted 2022-06-06; First posted 2022-06-10 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-05

CONDITIONS: Unplanned Hospital Readmissions; Patients at High Risk of Unplanned Readmission

STUDY DESIGN:
Intervention Model Description: intervention group (IG) or control group (CG). The IG will consist of placing the Epic 30-day unplanned readmission risk score in the story board of providers. If a patient is identified as having a high risk of readmission defined as readmission risk >20%, a link to transitional and supportive care services (TSC) will be appear in the story board. Providers will determine which TSC is best for the patient and may order whichever TSC or any is appropriate for the patient. The CG will have the same TSC orders available to them; however, they will not have the risk of readmission score present in their workflow, as such the embedded link to TSC will also not be present. Providers, in both IG and CG, will have the option to order one or multiple TSC at their discretion.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (IG) (Experimental): The IG will consist of placing the Epic 30-day unplanned readmission risk score in the story board of providers - If a patient is identified as having a high risk of readmission defined as readmission risk >20%, a link to transitional and supportive care services (TSC) will be appear in the story board
  Interventions: Behavioral: Epic 30-day unplanned readmission risk score
- control group (CG) (No Intervention): The CG will have the same transitional and supportive care services (TSC) orders available to them; however, they will not have the risk of readmission score present in their workflow

INTERVENTIONS:
Behavioral: Epic 30-day unplanned readmission risk score — If a patient is identified as having a high risk of readmission defined as readmission risk >20%, a link to transitional and supportive care services (TSC) will be appear in the story board.
  Arms: intervention group (IG)

SUMMARY:
The objective is to assess the implementation of a computerized clinical decision support (cCDS) tool for identifying patients at high risk of unplanned readmission who could benefit from existing care programs aimed at reducing readmissions

DETAILED DESCRIPTION:
Providers from either service, which includes attending physicians, residents, hospitalists, and advanced practice providers (APPs), will be randomly allocated to an intervention group (IG) or control group (CG). The IG will consist of placing the Epic 30-day unplanned readmission risk score in the story board of providers. If a patient is identified as having a high risk of readmission defined as readmission risk >20%, a link to transitional and supportive care services (TSC) will be appear in the story board. Providers will determine which TSC is best for the patient and may order whichever TSC is appropriate for the patient. The study team will not recommend TSCs. The risk of readmission score will be present from the time of admission for those in the IG. The CG will have the same TSC orders available to them; however, they will not have the risk of readmission score present in their workflow, as such the embedded link to TSC will also not be present.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Atrium Health Wake Forest Baptist Hospital (AHWFBH)
* 18 years or older
* meeting inpatient criteria
* admitted to hospitalist or general medicine teaching services
* Providers on the hospitalist or general medicine teaching services

Exclusion Criteria:

* Psychiatric diagnoses during index or subsequent admission
* left Against Medical Advice (AMA)
* planned readmission
* died during index admission
* Providers who opt out of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group
Number of transitional and supportive care services (TSC) referrals by providers in the Control group | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Faith Health | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Faith Health
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - High Risk Readmission Program (HRI) | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - High Risk Readmission Program (HRI)
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Care Plus | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Care Plus
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Population Health Pharmacy | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Population Health Pharmacy
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Geriatrics Transitional Care | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Geriatrics Transitional Care
Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Mobile Health Clinic | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Control group - Mobile Health Clinic
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Faith Health | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Faith Health
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group- High Risk Readmission Program (HRI) | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - High Risk Readmission Program (HRI)
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Care Plus | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Care Plus
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Population Health Pharmacy | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Population Health Pharmacy
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Geriatrics Transitional Care | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Geriatrics Transitional Care
Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Mobile Health Clinic | Day 30
  Number of transitional and supportive care services (TSC) referrals by providers in the Intervention group - Mobile Health Clinic
Provider Satisfaction Score | Day 30
  Provider satisfaction with clinical decision support tool measured by survey

SECONDARY OUTCOMES:
30 day Readmission Rate | Day 30
  proportion of index inpatient visits with an inpatient readmission within 30 days of index discharge

CONTACTS AND LOCATIONS:
Overall Officials: Donna Williams, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol Statistical Analysis Plan (SAP) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose